CLINICAL TRIAL: NCT03668405
Title: Interventional, Open-label, Multiple-immunization Extension Study on the Safety, Tolerability and Immunogenicity of Lu AF20513/Adjuvant in Patients With Alzheimer's Disease
Brief Title: A Study to Evaluate the Long-term Safety and Tolerability of Lu AF20513 and the Antibody Response in Patients With Alzheimer's Disease (AD)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: New data: The study was terminated based on new efficacy data from another study
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16026B; 2014-001797-34 (EudraCT Number)
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lu AF20513 high dose (Experimental)
  Interventions: Drug: Lu AF20513

INTERVENTIONS:
Drug: Lu AF20513 — Injection

SUMMARY:
The purpose of this study is to evaluate the long-term safety, tolerability and antibody response of Lu AF20513 in patients with Alzheimer's disease who have completed the 16026A study.

ELIGIBILITY:
Main inclusion criteria:

* The patient has completed the 16026A study and has received the last study treatment within 12 months of the screening visit for the present study.
* The patient has an MRI scan done in relation to study 16026A performed within 9 months before first study visit in the extension study.
* The patient has a knowledgeable and reliable caregiver/ study partner who will be available and able to accompany the patient to clinical visits, monitor Immunisation-Related Events after each immunisation, and participate with the patient at phone visits during the study

Main exclusion criteria:

* The patient uses or has recently used (pre-trial time limits specified in Appendix II) disallowed concomitant medication or it is anticipated that the patient will require treatment with at least one of the disallowed concomitant medications (Appendix II) during the study.
* The patient has a disease or takes medication that, in the opinion of the investigator, could interfere with the assessments of safety and tolerability

More inclusion and exclusion criteria may apply

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Baseline to week 96
  Based on the safety assessments (clinical safety laboratory tests, vital signs, ECGs, physical examinations (including neurological), Immunisation-Related Events (IRE) (selected from Brighton Collaboration guidelines) and magnetic resonance imaging (MRI) safety scans)
Aβ-specific antibody titre in plasma | Baseline to week 96

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (4):
- FI001, Turku, Finland
- Sweden (3):
  - SE002, Malmo
  - SE003, Mölndal
  - SE001, Stockholm